CLINICAL TRIAL: NCT00794859
Title: Trial of Sorafenib in Malignant Mesothelioma Previously Treated With Platinum-based Chemotherapy
Brief Title: Sorafenib in Previously Treated Malignant Mesothelioma
Acronym: SMS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Collaborators: Bayer (Industry)
Responsible Party: James Spicer, King's College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-005091-13
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sorafenib — 400mg twice daily

SUMMARY:
The principal objective of the study is to investigate the effect of sorafenib on progression free survival (time until the cancer begins to grow again,) in patients with malignant mesothelioma who have had prior treatment with chemotherapy. Effectiveness of the drug will also be explored with PET scans before and during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Malignant pleural or peritoneal mesothelioma previously treated with first line platinum-based chemotherapy (prior pemetrexed not required)
* Not suitable for radical resection. Prior radical or cytoreductive surgery allowed
* Age >18 years
* ECOG performance status 0-2
* Measurable disease. Lesions must be measured by CT scan or MRI according to modified RECIST (Appendix B)
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to start of first dose:

  * haemoglobin ≥ 9.0 g/dL
  * neutrophil count ≥ 1.5 x109/L
  * platelet count ≥ 100 x109/L
  * total bilirubin ≤ 1.5 x upper limit of normal
  * ALT and AST ≤ 2.5 x upper limit of normal (≤ 5 x upper limit of normal for *alkaline phosphatase ≤ 4 x upper limit of normal
  * PT-INR (international normalized ratio of PT) / PTT ≤1.5 x upper limit of normal
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to performing any study specific procedures.

Exclusion Criteria:

* History of cardiac disease: congestive heart failure > NYHA (New York Heart Association) class 2; active coronary artery disease (myocardial infarction more than 6 months prior to study entry is allowed); cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted); or uncontrolled hypertension (defined as systolic blood pressure >150mmHg or diastolic pressure >90mmHg despite optimal medical management)
* Impaired immunity or chronic infection including history of HIV (human immunodeficiency virus) infection or chronic hepatitis B or C
* Active clinically serious infections (> grade 2 NCI-CTCAE version 3.0)
* Seizure disorder requiring medication (such as steroids or anti-epileptics)
* Known brain metastasis. Patients with neurological symptoms should undergo a CT scan/MRI of the brain to exclude brain metastasis
* History of organ allograft
* Evidence or history of bleeding diathesis or coagulopathy;
* Renal dialysis
* Cancer other than mesothelioma within 5 years prior to start of study treatment EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, or superficial bladder tumours [Ta (noninvasive tumour), Tis (carcinoma in situ) & T1 (tumour invading lamina propria)]
* Thrombotic or embolic events such as cerebrovascular accident including transient ischemic attacks within the past 6 months
* Pulmonary haemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug
* Any other haemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug
* Serious, non-healing wound, ulcer, or bone fracture
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate birth control measures during the course of the trial. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Any condition that is unstable or could jeopardise the safety of the patient and their compliance in the study
* Patients unable to swallow oral medications
* Any malabsorption condition.
* Any prior systemic anticancer therapy including cytotoxic therapy, targeted agents, experimental therapy, adjuvant, or neo-adjuvant therapy for malignant mesothelioma, other than first line platinum-based combination chemotherapy
* Radiotherapy during study or within 3 weeks of start of study drug. (Palliative radiotherapy will be allowed as described in the Prior and Concomitant Therapy section)
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first dose of study drug (bronchoscopy is allowed)
* Granulocyte colony stimulating factor (GCSF) or granulocyte macrophage colony stimulating factor (GMCSF), within 3 weeks of study entry
* Therapeutic anticoagulation with vitamin K antagonists such as warfarin, or with heparins or heparinoids. Low dose warfarin (1 mg po OD) is permitted if the INR (international normalized ratio) is < 1.5. Low-dose aspirin is permitted (≤ 81 mg daily)
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 24 weeks

SECONDARY OUTCOMES:
Response rate as assessed with CT scan | 2 months
Overall survival | Median
Change in FDG-PET avidity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James Spicer, MRCP, PhD, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom